CLINICAL TRIAL: NCT05015725
Title: A Single Center Cross-sectional Study to Evaluate the Relationship Between Serum rT3 Concentrations, T3/T4 Ratio, and Symptoms/Quality of Life in Treated Hypothyroid Patients
Brief Title: The Relationship Between Serum rT3 Concentrations, T3/T4 Ratio, and Symptoms/Quality of Life in Treated Hypothyroid Patients
Status: Completed | Type: Observational
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Istvan Takacs, Director of Department, Semmelweis University
Other Study IDs: RT3QoLSE
Record Dates: First submitted 2021-06-30; First posted 2021-08-20 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Hypothyroidism
Keywords: hypothyroidism; reverse T3; quality of life
MeSH Terms: conditions — Hypothyroidism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treated hypothyroidism: Patients with treated hypothyroidism
  Interventions: Diagnostic Test: Quality of life assessment, biochemical measures

INTERVENTIONS:
Diagnostic Test: Quality of life assessment, biochemical measures — Psychological tests: ThyDQol, ThySRQ and the Somatosensory Amplification Scale (SASS) adding up to ~50 items including demographic variables.
  Recording of basic anthropometric data. Blood draw Laboratory tests: TSH, T3, FT3, FT4, aTPO, rT3, serum cholesterol, CK, GOT, GPT, creatinine and sodium levels.

SUMMARY:
The aim of this study is to evaluate the relationship between serum rT3 (serum reverse triiodothyronine) concentrations, T3/T4 (triiodothyronine/thyroxine) ratio, and persistent symptoms /quality of life in treated hypothyroid patients.

Investigators are going to measure TSH (thyroid stimulating hormone), free-T3, free-T4, reverse-T3 levels, biochemical markers of hypothyroidism and quality of life (assessed by validated questionnaires).

DETAILED DESCRIPTION:
Rationale: L-thyroxin (T4) substitution is the mainstay of treatment for hypothyroidism irrespective of disease origin. In a subset of patients with hypothyroidism however an inadequate peripheral T4->T3 conversion is hypostasized by some authors. This is speculated to lead to tissue level hypothyroidism and persistent symptoms even with adequate T4 replacement. As a potential pathogenetic mechanism, the inborn or acquired defect of peripheral deiodinases, decreased T3 and increased rT3 production is suggested.

Few results support this hypothesis. A decreased T3/T4 ratio has been reported in some post-surgical hypothyroid patients, while a few studies patient show increased patient satisfaction with combined T4+T3 substitution. However these differences have not been shown to be significant in large meta-analyses.

Due to the lack of convincing evidence current guidelines advocate against both routine rT3 measurement and T3 substitution. However in recent years, rT3 measurement and T3 supplementation has been steadily gaining popularity amongst some medical and functional medicine practitioners. Recent publications estimate order volume for rT3 tests in the US to be over 1 million per year. Thus, despite several decades of experience and multiple trials, the role of liothyronine (T3) substitution remains somewhat controversial.

The relationship between rT3 levels, T3/T4 ratio, quality of life and persistent symptoms of hypothyroidism in patients treated with adequate thyroxine doses has not been previously assessed.

A significant association of this nature would suggest the possibility of decreased peripheral T4->T3 conversion in some patients leading to worse treatment outcomes. A lack of relationship would further discredit the above detailed theories and could potentially help reduce the inadequate use of T3 substitution in patients.

Study population: Patients treated for hypothyroidism with no significant comorbidities are to be enrolled. Sample size calculations show adequate statistical power with over 150 participants. Based on the number of hypothyroid patients at our outpatient clinic, a sample size of 300-350 patients can reasonably be expected.

Schedule of activities: All study related procedures are performed during a single visit. These include recording of basic anthropometric data, a single draw of blood, and administration of psychological questionnaires. Laboratory tests include comprehensive thyroid function testing (TSH, T3, FT3, FT4, aTPO [anti-thyroperoxidase antibody]) with the addition of rT3 measurement. Less specific markers, associated with hypothyroidism are also assessed. These include serum cholesterol, CK (creatin-kinase), GOT/ASAT (aspartate-aminotransferase), GPT/ALAT (alanine-aminotransferase), creatinine and sodium levels. Psychological tests administered at the visit include ThyDQol, ThySRQ and the Somatosensory Amplification Scale (SASS) adding up to ~50 items including demographic variables.

Statistical analysis: Statistical methods for this study possibly include correlation analysis, linear and logistic regression.

Objectives and endpoints: Current understanding of hypothyroidism and thyroid hormone replacement imply that treatment with thyroxine doses that are sufficient to the normalize TSH lead to adequate tissue T3 levels and euthyroid state in the whole body. An association however between quality of life and rT3, levels or T3/T4 ratio could point out patients that could potentially benefit from additional T3 replacement.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age, inclusive, at the time of signing informed consent form.
* Hypothyroidism treated for >2 years
* TSH stable between 0.4 and 4.0 mIU/L for the past 6 months (at least 2 measurements)

Exclusion Criteria:

* Abnormal TSH on screening
* Unwilling or unable to participate/sign informed consent
* Changes in thyroxine dose or any other medication in the previous month
* Severe obesity (BMI [body mass index] >35kg/m2)
* Other significant comorbidity:
* History of ischaemic heart disease, valvular defect, stent placement, heart failure, stroke or TIA (transient ischemic attack)
* Diabetes mellitus under OAD (oral antidiabetic drug) or insulin treatment
* eGFR (estimated glomerular filtration rate) <60ml/min at screening, calculated by EPI formula
* History of liver disease, AST/ALT>3 times normal or GGT (gamma-glutamil transferase) >2 times normal or hyperbilirubinaemia at screening
* Systemic autoimmune condition currently under treatment (RA [rheumatoid arthritis], lupus, systemic sclerosis etc.)
* Active malignancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients treated for hypothyroidism with levothyroxine substitution.
Sampling Method: Non-Probability Sample
Enrollment: 262 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Association between rT3 level and quality of life | baseline
  Result of linear regression for evaluating the possible relation between serum reverse-T3 level and quality of life (QoL). For QoL assessment we are going to use the total points achieved on ThyDQol, ThySRQ and the Somatosensory Amplification Scale (SASS) tests.
Association between rT3 level and SASS result | baseline
  Result of linear regression for evaluating the possible relation between serum reverse-T3 level and the result of Somatosensory Amplification Scale (SASS) questionnaire.
Association between rT3 level and ThySRQ result | baseline
  Result of linear regression for evaluating the possible relation between serum reverse-T3 level and the result of ThySRQ questionnaire.
Association between rT3 level and ThyDQol result | baseline
  Result of linear regression for evaluating the possible relation between serum reverse-T3 level and the result of ThyDQol questionnaire.

SECONDARY OUTCOMES:
Association between rT3 and LDL-cholesterol level | baseline
  Result of linear regression for evaluating the possible relation between serum reverse-T3 and LDL-cholesterol level.
Association between rT3 and CK level | baseline
  Result of linear regression for evaluating the possible relation between serum reverse-T3 and creatin-kinase level.
Association between rT3 and GOT/ASAT level | baseline
  Result of linear regression for evaluating the possible relation between serum reverse-T3 and GOT/ASAT level.
Association between rT3 and GPT/ALAT level | baseline
  Result of linear regression for evaluating the possible relation between serum reverse-T3 and GPT/ALAT level.
Association between rT3 and eGFR level | baseline
  Result of linear regression for evaluating the possible relation between serum reverse-T3 and eGFR level (eGFR will be calculated by using EPI formula).
Association between rT3 and sodium level | baseline
  Result of linear regression for evaluating the possible relation between serum reverse-T3 and sodium level.

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University - Departement Medicine and Oncology, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No